CLINICAL TRIAL: NCT07362017
Title: A Multicenter, Open Label Study to Investigate the Safety and Efficacy of Ponesimod in the Treatment of Moderate-to-Severe Chronic Plaque Psoriasis
Brief Title: Open Label Study to Investigate the Safety and Efficacy of Ponesimod in Moderate-to-Severe Chronic Plaque Psoriasis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-VSP-128-3102
Record Dates: First submitted 2026-01-20; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Moderate-to-severe Chronic Plaque Psoriasis
Keywords: psoriasis; Moderate-to-severe chronic plaque psoriasis
MeSH Terms: conditions — Psoriasis | interventions — ponesimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ponesimod (Experimental): Ponesimod
  Interventions: Drug: Ponesimod

INTERVENTIONS:
Drug: Ponesimod — Oral Tablet

SUMMARY:
An open label study to investigate the safety and efficacy of ponesimod in participants with moderate-to-severe chronic plaque psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18-65 years, inclusive
* BMI >18 and <40
* Minimum affected BSA of 10%
* PASI score ≥ 12
* PGA ≥ 3
* Diagnosed with moderate-to-severe plaque psoriasis

Exclusion Criteria:

* Diagnosis of generalized erythrodermic, generalized pustular (von Zumbusch), guttate, or palmoplantar psoriasis
* History of an allergic reaction or known and/or significant sensitivity to study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of ponesimod as measured by reporting of adverse events (AEs) | Through study completion, approximately 1 year
  Safety will be assessed based on frequency of treatment-emergent adverse events and serious adverse events, and frequency of clinically notable abnormal vital signs, blood chemistry, hematology, urology, and ECGs

IPD SHARING:
Plan to Share IPD: No